CLINICAL TRIAL: NCT06593795
Title: Prediction of External Cephalic Version Success in Case of Breech Presentation At Term of Pregnancy: a Prospective Observational Study
Brief Title: Ultrasound Parameters for the Outcome Prediction of External Cephalic Version for Fetuses with Breech Presentation
Acronym: REVERSO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Carducci Brigida, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6366
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Breech Fetal Presentation; Breech Presentation of Fetus with Successful Version; Vaginal Delivery; Cesarean Section
Keywords: breech; external cephalic version; ultrasound; c-section
MeSH Terms: conditions — Breech Presentation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group ECV: Pregnant women with a fetus in breech presentation at term of pregnancy undergoing an external cephalic version (ECV) maneuver. This procedure is aimed to induce fetal cephalic position allowing vaginal delivery instead of cesarean section
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — before ECV procedure, an ultrasound will be performed to evaluate
  * fetal biometry (BPD, HC, AC, FL, EFW);
  * Occiput position (right, left);
  * Back position (anterior, posterior, right, left);
  * Breech variant (footling, frank, complete);
  * Fetal leg posture (extended, flexed)
  * Placental localization;
  * Amniotic Fluid Index (AFI);
  * Fore-bag of amniotic fluid;
  * Eventual presence of nuchal cords;
  * Fetal head ballottement (yes, no);
  * Occiput-spine angle These parameters will be compared to find predictive factors for successful ECV

SUMMARY:
This study aims to evaluate possible predictors for the successful od external cephalic version (ECV), a procedure that is indicated in your case due to breech presentation of your baby and your desire to avoid cesarean section. Before the procedure, a detailed ultrasound scan will be performed to measure several parameters. After the procedure we will collect data about the duration, outcome and eventual complications of ECV.

DETAILED DESCRIPTION:
Pregnant women with a diagnosis of fetal breech presentation, desirous of an attempt of ECV after counseling and written consent and hospitalized for the procedure will be consecutively enrolled. The following anonymous data will be recorded:

* Demographic and anthropometric data (i.e., age (y), ethnicity, height (m), weight (kg), BMI);
* Parity
* Gestational Age (weeks + days)

Before ECV attempt, the following evaluations will be performed:

* Vaginal examination to evaluate the cervical dilatation and the level of presenting part (floating or not floating)
* Fetal transvaginal ultrasound reporting:

  * biometry (BPD, HC, AC, FL, EFW);
  * Occiput position (right, left);
  * Back position (anterior, posterior, right, left);
  * Breech variant (footling, frank, complete);
  * Fetal leg posture (extended, flexed)
  * Placental localization;
  * Amniotic Fluid Index (AFI);
  * Fore-bag of amniotic fluid;
  * Eventual presence of nuchal cords;
  * Fetal head ballottement (yes, no);
  * Occiput-spine angle (see Figure 1)

Then, all the participants will undergo a transabdominal ultrasound-guided ECV in a semi-sitting position by the same expert operator (B.C.). After the procedure, the following data will be collected:

* Success (yes, no)
* Duration of the procedure (min);
* Direction of fetal flip in case of success (frontside flip, backside flip)
* Pain perception in Numerical Rating Scale (NRS) (1-10);
* Reason for terminating the procedure (success, failure, pain, uterine contractions, non-reassuring fetal conditions)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 y.o.;
* Pregnant women with a diagnosis of fetal breech presentation eligible and desirous for ECV;
* Singleton;
* At term (≥ 37 weeks);
* Breech presentation;
* No previous uterine scars or other indications for elective C-section;
* Signed written informed consent to study participation.

Exclusion Criteria:

* Age <18 y.o.;
* Preterm gestational age;
* Multiple pregnancies;
* Indications for elective cesarean section;
* Incomplete obstetrical data;
* Refusal to provide informed consent.
* Desire to an elective C-Section
* Controindications for ECV or vaginal delivery (placental abruption, placenta previa, uterine malformations)
* Reduction of amniotic fluid (AFI <4 cm)
* Uterine contractions
* Vaginal bleeding
* Premature rupture of membranes
* Nonreassuring fetal heart rate patterns before the procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will consecutively enroll all pregnant women at the term of gestation with a fetal breech presentation undergoing ECV attempt after counseling at Fondazione Policlinico Universitario Agostino Gemelli IRCCS of Rome, satisfying the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate ECV success rate. | during the procedure
  to evaluate clinical and ultrasound parameters possibly predictive of the success of ECV. This will allow the creation of a predictive model for adequate counseling for the women undergoing the procedure for the cephalic version of fetuses in breech presentation at term of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: silvio tartaglia, MD, Study Director — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No
this is an internal database